CLINICAL TRIAL: NCT02857959
Title: Doctor of Medicine
Brief Title: One Dose Versus Three Weekly Doses of Benzathine Penicillin G for Patients With Early Syphilis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jun Li (Other)
Responsible Party: Sponsor-Investigator, Jun Li, M.D., Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PUMCH-2016078
Record Dates: First submitted 2016-08-03; First posted 2016-08-05 (Estimated); Last update posted 2018-11-16 (Actual); Status verified 2018-11

CONDITIONS: Syphilis
MeSH Terms: conditions — Syphilis | interventions — Penicillin G

ARMS (2):
- single dose benzathine penicillin G. (Experimental): single dose benzathine penicillin G.
  Interventions: Drug: Benzathine Penicillin G
- three doses of benzathine penicillin G. (Active Comparator): three doses of benzathine penicillin G.
  Interventions: Drug: Benzathine Penicillin G

INTERVENTIONS:
Drug: Benzathine Penicillin G

SUMMARY:
The purpose of this study is to observe the serological response to 1 or 3 weekly doses of benzathine penicillin G in patients with early syphilis.

ELIGIBILITY:
Inclusion Criteria:

1. Persons with confirmed early symptomatic syphilis (primary or secondary) or high-titer latent syphilis
2. A rapid plasma reagin (RPR) test was positive, with a titer were 1:4 or higher. In addition, Treponema pallidum particle agglutination assay and/or fluorescent treponemal antibody absorption test were reactive.

Exclusion Criteria:

1.Patients who were pregnancy, known allergy to penicillin, use of antibiotics active against syphilis during the preceding six months for symptomatic cases or during the preceding two years for asymptomatic cases, and concurrent illnesses requiring treatment with antibiotics effective against syphilis. 2. if RPR titers were found to be 1:4 or less or the T. pallidum particle agglutination test was nonreactive, participants were retrospectively excluded from the trial unless primary syphilis was confirmed by the finding of T. pallidum in ulcer exudates on direct immunofluorescence

-

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-08; Primary Completion 2020-06 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Rapid plasma reagin titers | up to 9 months after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Dermatology and Venereology, Peking Union Medical College Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, China, Beijing, China